CLINICAL TRIAL: NCT00578084
Title: Lung Cancer Location: A Prospective Repository
Brief Title: Lung Cancer Location: a Repository
Status: Terminated | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 0604-76; IRB # 0604-76
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- surgery: those subjects who went to surgery to treat their lung cancer
- no surgery: those subjects who did not go to surgery for their lung cancer
- NSCLC: subjects with NSCLC
- Small cell lung cancer: those with small cell lung cancer

SUMMARY:
The purpose of this repository is to prospectively examine subjects with known or suspected lung cancer to determine the extent of mediastinal lymph node involvement with respect to primary lung cancer location. The data collected in this repository may be used to influence our current standard of care and streamline indications for EUS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing EUS evaluation of a mediastinal mass, or suspected/known lung cancer
* Subjects with a prior history of lung cancer
* Subjects referred to thoracic surgery for evaluation of a suspected/known lung cancer

Exclusion Criteria:

* Altered mental status that would prohibit the giving and understanding of informed consent
* Dementia
* Psychiatric illness that would preclude adequate compliance with communication for this protocol
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with known or suspected lung cancer will be identified by referral to the thoracic surgeon or ultrasonographer at the Veterans Affairs Hospital or Indiana University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
examine subjects with known or suspected lung cancer to determine the extent of mediastinal lymph node involvement with respect to primary lung cancer location | ongoing-database

CONTACTS AND LOCATIONS:
Overall Officials: Julia LeBlanc, MD, MPH, Principal Investigator — Indiana University
Locations (1):
- Clarian/IUPUI: University Hospital, Indianapolis, Indiana, United States